CLINICAL TRIAL: NCT03407183
Title: The Efficacy of Botulinum Toxin in Spastic Neuropathic Bladder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: AHMED FARAHAT HASSAN (Other)
Responsible Party: Sponsor-Investigator, AHMED FARAHAT HASSAN, Principal Investigator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: botox in neurogenic bladder
Record Dates: First submitted 2017-12-29; First posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Spastic Neurogenic Bladder
MeSH Terms: conditions — Urinary Bladder, Neurogenic | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- spastic neurogenic bladder: intradetrusor injection of botulinumtoxinA (Botox®, Allergan, Irvine, USA) in patients with spastic neurogenic bladder is 200 U of onabotulinumtoxinA once, then follow up after three months.
  Interventions: Procedure: intradetrusor injection of botulinumtoxinA (Botox)

INTERVENTIONS:
Procedure: intradetrusor injection of botulinumtoxinA (Botox) — intradetrusor injection of botulinumtoxinA (Botox®, Allergan, Irvine, USA) to assess the efficacy of Botox in treatment of neurogenic bladder.

SUMMARY:
To assess the efficacy of botulinum toxin in spastic neurogenic bladder.

DETAILED DESCRIPTION:
Neurogenic detrusor overactivity (NDO) can result in lower and upper urinary tract complications and eventually even in end-stage kidney failure. Since the driving force of this clinical cascade is high bladder pressure, controlling intravesical pressure in NDO patients improves both quality of life and life-expectancy in these patients. Botulinum toxin A (BTX-A) has proven its efficacy in reducing intravesical pressure and in reducing incontinence episodes. BTX-A also improves quality of life in patients with NDO. Both onabotulinumtoxinA (Botox®, Allergan, Irvine, USA) and abobotulinumtoxinA (Dysport®, Ipsen, Paris, France) have a level A recommendation for NDO-treatment. The recommended dose for intradetrusor injections in NDO patients is 200 U of onabotulinumtoxinA or 500 U of abobotulinumtoxinA. The drug is generally administered extratrigonal in the detrusor muscle, via cystoscopic guided injection at 20 sites in 1 mL injections. Intradetrusor BTX-A injections are safe, with mostly local complications such as urinary tract infection and high post-void residual or retention. The effect of the toxin lasts for approximately 9 months. Repeat injections can be performed without loss of efficacy. Different injection techniques, novel ways of BTX-A administration, eliminating the need for injection or new BTX-A types with better/longer response rates could change the field in the future.

Botulinum toxins are neurotoxins produced by the facultative anaerobe Clostridium botulinum that block the release of acetylcholine into the synaptic gap of the neuromuscular junction. Their injection near the nerves that supply the target organ selectively and temporarily paralyzes the organ. In particular, the subtype botulinum-A toxin is widely used in neurology to release spastic dystonia in adults and children . In urologic disorders, botulinum-A toxin reliably diminishes external sphincter or detrusor overactivity.

ELIGIBILITY:
Inclusion Criteria:

-1- patients with spastic neurogenic bladder due to upper motor neuron lesion as (spinal cord lesions ,multiple sclerosis ,strokes,parkinsonism...........).

2- patients with spastic neurogenic bladder diagnosed clinically and urodynamically.

Exclusion Criteria:

* 1-patients with associated lower motor neuron lesions. 2-atonic bladder. 3-patients with diabetes mellitus.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with spastic neurogenic bladder will be diagnosed clinically and urodynamically with preoperative assessment through:
  .History. .Examination. .Urine analysis. .Abdominal ultrasound (to assess upper urinary tract and post micturation residual).
  .Kidney function tests. .Urodynamic study. The patients will be re evaluated after 3 months post botulinum toxin injection regarding to previous items.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-02-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
The Efficacy of Botulinum Toxin in Spastic Neuropathic Bladder | 1 year
  By improvement of symptoms and evaluation of urodynamic studies, Kidney function tests , abdominal ultrasound and urine analysis compared to preoperative results.

CONTACTS AND LOCATIONS:
Overall Officials: AHMED FARAHAT, master, Principal Investigator — Assiut University
Locations (1):
- Ahmed Farahat, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Schurch B, Stohrer M, Kramer G, Schmid DM, Gaul G, Hauri D. Botulinum-A toxin for treating detrusor hyperreflexia in spinal cord injured patients: a new alternative to anticholinergic drugs? Preliminary results. J Urol. 2000 Sep;164(3 Pt 1):692-7. doi: 10.1097/00005392-200009010-00018. PMID 10953127
- [Background] Kirschner J, Berweck S, Mall V, Korinthenberg R, Heinen F. Botulinum toxin treatment in cerebral palsy: evidence for a new treatment option. J Neurol. 2001 Apr;248 Suppl 1:28-30. doi: 10.1007/pl00007815. PMID 11357236